CLINICAL TRIAL: NCT06673485
Title: The Effect of Vitamin D and Calcium Supplement on Overall Body Bone Density and Implant Stability in Posterior Maxilla: a Randomized Clinical Trial
Brief Title: The Effect of Vitamin D and Calcium Supplement on Overall Body Bone Density and Implant Stability in Posterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mostafa Sharkawy, Resident at Oral and Maxillofacial Surgery, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AUAREC20210100-06
Record Dates: First submitted 2024-10-13; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Dental Implant
Keywords: maxillary sinus augmentation; Sinus graft; Internal Sinus lifting; Allogenic bone graft

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A : Patients received vitamin D and calcium supplementation during the healing period (Experimental): 1. Monthly intramuscular injections of vitamin D3 (300,000 I.U.) for three months, concurrent with six months of oral Maxical vitamin D supplementation post-implant placement.
  2. Daily intake of Maxical calcium carbonate tablets (600 mg elemental calcium) for six months.
  Interventions: Procedure: Patients received vitamin D and calcium supplementation during the healing period
- Group B: Patients have not received any nutritional supplementation during the healing period. (Experimental)
  Interventions: Procedure: Patients have not received any nutritional supplementation during the healing period.

INTERVENTIONS:
Procedure: Patients received vitamin D and calcium supplementation during the healing period — The proposed implant site and adjacent tissues were disinfected using betadine mouthwash, and standard infiltration anesthesia was administered both buccally and palatally. A paracrestal incision was then made over the intended implant location, and the mucoperiosteal flap was elevated to expose the underlying bone. Subsequently, an osteotomy was prepared using a 2.0 mm pilot drill, maintaining irrigation with sterile saline. The osseodensification protocol was employed with Densah burs in increasing diameters (2 mm, 3 mm, 4 mm) under copious irrigation. Throughout the osteotomy preparation, implant angulation was regularly checked using a paralling pin. Upon encountering haptic feedback, pressure was modulated to achieve the desired depth. The implant was then installed using a surgical handpiece, and the final insertion torque was recorded using a torque wrench, ensuring successful placement.
  During the healing period, the patients recieved Vitamin D and Calcium Supplements.
  Arms: Group A : Patients received vitamin D and calcium supplementation during the healing period
Procedure: Patients have not received any nutritional supplementation during the healing period. — The proposed implant site and adjacent tissues were disinfected using betadine mouthwash, and standard infiltration anesthesia was administered both buccally and palatally. A paracrestal incision was then made over the intended implant location, and the mucoperiosteal flap was elevated to expose the underlying bone. Subsequently, an osteotomy was prepared using a 2.0 mm pilot drill while maintaining irrigation with sterile saline. The osseodensification protocol was employed with Densah burs in increasing diameters (2 mm, 3 mm, 4 mm) under copious irrigation. Throughout the osteotomy preparation, implant angulation was regularly checked using a paraling pin. Upon encountering haptic feedback, pressure was modulated to achieve the desired depth. The implant was then installed using a surgical handpiece, and the final insertion torque was recorded using a torque wrench, ensuring successful placement. During the healing period, the patients did not receive vitamin or calcium supplements.
  Arms: Group B: Patients have not received any nutritional supplementation during the healing period.

SUMMARY:
The aim of the study is to evaluate the effect of Vit D and Calcium administration on allogragt bone maturation radiographically and histomorphometercally in maxillary sinus augmentation in cases of D4 bone density.

ELIGIBILITY:
Inclusion Criteria:

* Patient with residual bone height from 5 : 8 .
* Patient with insufficient Vit D levels.
* Patient with D4 bone density.

Exclusion Criteria:

* Patients that have aproporiate amount of Ca and Vit D.
* Sinus pathology that precludes routine sinus augmentation.
* Heavy smookers patients.
* Systemic diseases that interfere with bone maturion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-02 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The Implant Stability Quotient | Immediate post-operative, and 6 Months post-operative
  The Implant Stability Quotient (ISQ) will be assessed using the Osstell device, which provides a stability score ranging from 0 ISQ to 100 ISQ. Higher ISQ values indicate greater implant stability, with 0 ISQ representing the lowest stability and 100 ISQ the highest. This measure allows for consistent, objective assessment of implant stability across time points.

SECONDARY OUTCOMES:
DXA Scan | pre-operative, and 6 Months post-operative
  DXA scan was carried out to T-score. minimum is - 4 and maximum is 1. the more T-score, the better the bone density.
Vitamin D serum levels | Pre-operative, and 6 Months post-operative
  Vitamin D serum levels (nanograms per milliliter (ng/ml)) will be represented as values, with higher values indicating a better vitamin D status. This measurement provides an objective assessment of vitamin D levels across participants.
Calcium Serum Level | Pre-operative, and 6 Months post-operative
  Calcium serum levels (milligrams per deciliter (mg/dl)) will be measured, with higher values indicating better calcium status within the physiological range. This measurement provides an objective assessment of calcium levels across participants, allowing for consistent evaluation of calcium status.

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar University, Asyut, Egypt